CLINICAL TRIAL: NCT06426121
Title: Clinical Validation of BACTEC™ Plus Aerobic/F Culture Vials Compared With Equivalent Product
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: IDS-23CNBAC01
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- BD BACTEC™ Plus Aerobic/F Culture Vials(test): Additional blood sample collected compared to clinical routine care
  Interventions: Diagnostic Test: test Aerobic/F Culture Vials
- BD BACTEC™ Plus Aerobic/F Culture Vials(control): clinical routine care
  Interventions: Diagnostic Test: control Aerobic/F Culture Vials

INTERVENTIONS:
Diagnostic Test: test Aerobic/F Culture Vials — an additional blood sample will be collected compared to clinical routine of blood culture, inoculated into the test culture vial, and compared with the blood culture results of the control vial collected from the same site and the same puncture point
  Groups: BD BACTEC™ Plus Aerobic/F Culture Vials(test)
Diagnostic Test: control Aerobic/F Culture Vials — according to the clinical routine of blood culture, this blood sample should be collected and inoculated into the control vial, and its culture result will be collected
  Groups: BD BACTEC™ Plus Aerobic/F Culture Vials(control)

SUMMARY:
This study is a multi-center, randomized clinical validation. Subjects should be fully informed of this protocol and related risks, and can only be enrolled into this study after signing the informed consent form. Blood collection of the subjects at the same puncture point at a single site will be injected into the test vial and the control vial respectively, and the vials will be transferred to the BACTEC system for culture and the results will be observed. After the BACTEC system incubation completion, the vials will be subcultured. Strains grown on plates will be identified using appropriate methods and, if possible, at the species level.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to provide written informed consent to sponsor.
* Blood specimens
* Patients with suspected blood infection that have one or more of the following characteristics :

  a) Body temperature > 38°C or body temperature <36°C; b) chills; c) increased peripheral blood leukocyte count (count > 10.0×109/L, especially if there is a "left shift") or decrease (count < 3.0×109/L); d) Respiratory rate > 20 beats/min or arterial partial pressure of carbon dioxide (PaCO2) <32mmHg; e) Heart rate> 90 beats/min; f) mucocutaneous hemorrhage; g) coma; h) Multi-organ dysfunction; i) decreased blood pressure; j) Elevated inflammatory response parameters such as C-reactive protein or hypersensitive C-reactive protein, procalcitonin (PCT), 1,3-β-D-glucan (G test), etc.

Exclusion Criteria:

* Subjects have been enrolled in this study and samples have been collected
* Patients with severe and very severe anemia (last hemoglobin <60g/L within seven days)
* Females with known pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with suspected blood infection who are at risk of sepsis
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
consistency rate | 8 days
  The consistency rate of the test vials and the control vials BACTEC™ system test results, including the overall consistency rate, positive consistency rate, and negative consistency rate

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No